CLINICAL TRIAL: NCT05581680
Title: Multimodal Quantified Analysis of Facial Movements: Comparison Between Pathological
Brief Title: Multimodal Quantified Analysis of Facial Movements: Comparison Between Pathological and Control Subjects
Acronym: AQ2MF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0207
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Electromyography; Eye-tracking; Facial Palsy
Keywords: facial mimics; motion capture; electromyography; eye-tracking; Facial Palsy
MeSH Terms: conditions — Facial Paralysis | interventions — Dental Impression Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with facial palsy (Experimental)
  Interventions: Other: dental impressions; Other: Simultaneous MoCap and EMG acquisition; Other: Eye-tracking acquisition for pathological subjects; Other: Follow-up visit for pathological subjects
- healthy volunteers (Active Comparator)
  Interventions: Other: dental impressions; Other: Simultaneous MoCap and EMG acquisition

INTERVENTIONS:
Other: dental impressions — dental impressions
Other: Simultaneous MoCap and EMG acquisition — Simultaneous MoCap and EMG acquisition
Other: Eye-tracking acquisition for pathological subjects — Eye-tracking acquisition for pathological subjects
  Arms: patients with facial palsy
Other: Follow-up visit for pathological subjects — Follow-up visit for pathological subjects
  Arms: patients with facial palsy

SUMMARY:
The facial palsy is a frequent disease with a lot of etiologies. It has variable severities with sometimes heavy functional repercussions and different recovery potentials. The proposed treatments are based on surgery, physiotherapy and botulinum toxin injections. However, when recovery is incomplete, acceptance is more difficult, with an impacted quality of life. Thanks to Motion Capture and Electromyography, a quantification of the facial mimicry is now possible with a great precision. In addition with the quantification of the facial mimicry, eye-tracking, wich is widely used in the marketing field, but it also finds medical applications including head and neck lesions and facial palsy in particular, will be used to evaluate the visio of the patients on their pathology in function of the movement quantification measured with MoCap and Electromyography. The aim of this research is to measure in a combined way the action potentials by sEMG and the amplitudes of displacement of the markers in motion capture, for movements determined in a population of patients presenting a facial pathology, in order to compare them with reference values obtained in healthy subjects. In a second step, the aim will be to study if there is a link between the way the patient looks at his pathology and the results of his management (treatment, rehabilitation) which will be quantitatively evaluated thanks to MoCap and sEMG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no known facial pathology (healthy volunteers) OR
* Patients with peripheral facial palsy, irrespective of grade, whether or not previously treated
* Subject with written informed consent
* Subject over 18 years of age
* Subject affiliated to a social security scheme

Exclusion Criteria:

* Subjects with severe skin disorders that do not allow the application of electrodes or photo reflective markers
* Subjects with speech disorders making it impossible to pronounce the sounds [o] and [pu]
* Subject unable to provide written informed consent
* Subjects under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
determination of baseline values of facial mimicry (in millimetres) in healthy volunteers | one month
  determination of baseline values of facial mimicry (in millimetres) in healthy volunteers
determination of baseline values of eye-tracking (in millimetres) in healthy volunteers | one month
  determination of baseline values of eye-tracking (in millimetres) in healthy volunteers
determination of the maximum range of motion of facial mimicry (in millimetres) in patients | one year
  determination of the maximum range of motion facial mimicry (in millimetres) in patients
determination of the maximum range of motion of eye-tracking (in millimetres) in patients | one year
  determination of the maximum range of motion of eye-tracking (in millimetres) in patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No